CLINICAL TRIAL: NCT06675487
Title: Polish Adaptation and Validation of Questionnaires for Assessing the Functional Efficiency of the Upper Limb After Stroke.
Brief Title: Assessment of Functional Efficiency of the Upper Limb After Stroke
Status: Recruiting | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Krzysztof Bylicki, Principal Investigator, University of Rzeszow
Other Study IDs: 035/06/2024
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; Ischemic; Rehabilitation; functional efficiency
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study will be to: conduct the process of cultural and linguistic adaptation of questionnaires for assessing the functional efficiency of the upper limb to the Polish version and to assess psychometric properties: reliability, validity and sensitivity to clinical changes among patients after stroke.

DETAILED DESCRIPTION:
Conducting the process of cultural and linguistic adaptation of questionnaires to the Polish version and assessing psychometric properties: reliability, validity and sensitivity to clinical changes of questionnaires for assessing the functional efficiency of the upper limb among patients after stroke. The following questionnaires will be used:

* The Motor Activity Log (MAL) Rasch-Based MAL-18
* The Chedoke Arm and Hand Activity Inventory (CAHAI) -- D u r u ö z H a n d I n d e x ( D H I ) Internal and external consistency between questions (whether they are used to assess the same phenomenon/function) and studies will be conducted twice (first time, and then after 2 weeks by three researchers under the same conditions.

To assess the validity and sensitivity of the tools, patients will be additionally assessed:

* Barthel scale
* VAS scale
* WHOQOL-BREF questionnaire for assessing quality of life
* Stroke Quality of Life Scale - (SSQOL).
* Functional electrostimulation and EMG
* The Modified Ashworth Scale (MAS)
* Box and Blocks
* Franchay scale
* Fugl-Meyer Motor Assessment Scale for Upper Extremity
* measurement using a dynamometer and pinchmeter
* measurement using the R500 goniometer

After assessing the reliability and validity of the tools, the sensitivity will be assessed based on the assessment of the effects of rehabilitation in people after a stroke before the start of the stay and after the 3-week rehabilitation program.

Procedure for testing the sensitivity of the research tools:

The subjects will participate in a 3-week rehabilitation program from Monday to Friday, 15 days in the stay. Each patient staying at the spa hospital participated in a comprehensive rehabilitation program conducted during the day, lasting from 120 to 150 minutes.

The program will include: group and individual exercises (active, assisted, manipulation exercises, exercises using the PNF method, balance exercises, breathing exercises), manual massage, physical treatments such as: laser, whirlpool bath, mud compresses, carbon dioxide bath, tens currents, bio-v lamp, local cryotherapy, training with biofeedback aimed at improving the motor function of the hand. A Biometrics device will be used for the exercises. The device allows for movements in all planes of individual hand joints. During the exercises, the patient has a visualization of the movements he performs on the monitor screen, thanks to which he can influence the increase in the range of movement and engage greater muscle strength through biofeedback, additionally, the confirmation of correct performance of the task is a visual assessment. The duration of the exercises with the biofeedback function will be 30 minutes a day. Additionally, anthropometric measurements will be performed among the patients.

Body weight will be measured to the nearest 0.1 kg. The content of adipose tissue (FAT), lean tissue (FFM), muscle tissue (PMM), bone tissue (BM) and water (TBW) will be analyzed. Body mass components will be assessed on a Tanita MC 780 MA body composition analyzer using the bioelectrical impedance method (BIA).

Body height will be measured to the nearest 0.1 cm using a portable PORTSTAND 210 stadiometer. Measurements will be performed under standard conditions. For the study, each participant will stand upright under the supervision of the research team and with bare feet.

Body mass index (BMI) will be calculated by dividing the body mass (kg) of each individual by their body height squared (m2). After obtaining the results regarding height and weight, the body mass index (BMI) will be calculated, and then the BMI value will be related to the obesity classification according to the WHO: ≤ 18.49 underweight, 18.5 - 24.99 normal body weight, 25 - 29.99 overweight, ≥ 30 obesity.

The research will be conducted at the Spa and Rehabilitation Hospital in Iwonicz Zdrój. After meeting the inclusion criteria, qualification for the study will be performed. The internal and external reliability of the tools will be assessed twice (first time and then after 2 weeks by three researchers in the same conditions). Then the accuracy of the selection of tools will be assessed based on the selected scales, questionnaires.

After assessing the reliability and validity of the tools, sensitivity will be assessed based on the assessment of rehabilitation effects in people after stroke before the start of the stay and after the 3-week rehabilitation program. The study is planned to be conducted in the morning hours. The study time for one participant will be 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* informed, voluntary consent of the patient
* completed, single ischemic stroke
* hemiparesis
* time since stroke at least 6 months
* age 45-75 years
* elementary (basic) grip ability
* degree of paresis of the upper limb, hand and lower limb 4-5 on the Brunnström scale
* degree of disability on the Rankin scale 3
* spastic tone of the paretic upper limb, hand and lower limb no more than 1 plus on the modified Ashworth scale - current health condition confirmed by a medical examination allowing participation in the tests and exercises

Exclusion Criteria:

* lack of informed, voluntary consent of the patient

  * second or subsequent stroke, hemorrhagic stroke, stroke of the brain stem and cerebellum
  * disorders of higher mental functions limiting understanding and carrying out tasks during exercises
  * visual field disorders
  * mechanical and thermal injuries that may affect the limitation of the grip function of the hand
  * coexisting neurological, rheumatological, orthopedic diseases, including fixed contractures that may affect the grip ability and locomotion
  * unstable medical condition
* metal implants, electronic implants, menstruation in women, epilepsy,
* failure to complete a 3-week rehabilitation stay

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned group size is 100 patients with hemiparesis after stroke staying on a rehabilitation stay at the Excelsior Spa and Rehabilitation Hospital in Iwonicz Zdrój.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The Motor Activity Log (MAL) | Internal and external reliability of the tools: assessed twice (first time and then after 2 weeks). After assessing the reliability and validity of the tools, sensitivity will be assessed (before the start of the stay and after 3 weeks of rehabilitation)
  The Motor Activity Log (MAL) - a subjective scale, consisting in assessing the quantity and quality of movements of the directly affected limb, outside laboratory conditions. Participants of the study answer 30 standardized questions about the amount of movement (Amount Scale or AS) and quality of movement (How Well Scale or HW) in the directly affected limb. The scales are located on separately printed forms, the subjects are informed about the method of assessment, as well as the possibility of entering half-grades (e.g. 0.5, 4.5).
  Where 0 means that there is no possibility of movement and 5 means that the arm movement is possible.
Rasch-Based MAL-18 | Internal and external reliability of the tools: assessed twice (first time and then after 2 weeks). After assessing the reliability and validity of the tools, sensitivity will be assessed (before the start of the stay and after 3 weeks of rehabilitation)
  Rasch-Based MAL-18 - is a shortened version of MAL-28, the examined person answers questions about 18 actions (from simple to alternative, leading actions) and advises them in the following way: 0 points - ends not used 0 points - movement is in a very small size 0 points - movement ends with paralysis requires dependent assistance 1 point - movement ends in a height encompassing 2 points - movement almost within the norm 3 points - movement within the norm.
The Chedoke Arm and Hand Activity Inventory (CAHAI) | Internal and external reliability of the tools: assessed twice (first time and then after 2 weeks). After assessing the reliability and validity of the tools, sensitivity will be assessed (before the start of the stay and after 3 weeks of rehabilitation)
  Is used to assess upper limb function, consists of 13 activities that the examined person has to perform. Activity Scale:
  1. total assist (weak U/L < 25%)
  2. maximal assist (weak U/L = 25-49%)
  3. moderate assist (weak U/L = 50-74%)
  4. minimal assist (weak U/L > 75%)
  5. supervision
  6. modified independence (device)
  7. complete independence (timely, safely)
D u r u ö z H a n d I n d e x ( D H I ) | Internal and external reliability of the tools: assessed twice (first time and then after 2 weeks). After assessing the reliability and validity of the tools, sensitivity will be assessed (before the start of the stay and after 3 weeks of rehabilitation)
  18 questions regarding ability to carry out manual tasks. Questions are grouped in five domains: In the kitchen (8), dressing (2), hygiene (2), in the office (2), and other (4) The patient is instructed to answer each question in terms of the level of difficulty they experience completing various tasks without help from another person or assistive device (Sezer, Yavzer, Sivrioglu, Basaran, & Koseoglue, 2006) Individual items are scored on a 6-point Likert scale where 0=without difficulty and 5=impossible. The 18 individual scores are summed to obtain a composite score The total score ranges from 0-90 with higher scores indicating poorer hand functioning

SECONDARY OUTCOMES:
Barthel scale | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Barthel scale - to assess activities of daily living. A maximum of 100 points can be obtained. Based on the points awarded, we assess the patient's condition as: I. 86-100 points - patient's condition "mild"; II. 21- 85 points - patient's condition "moderately severe"; III. 0 - 20 points - patient's condition "very severe".
VAS scale | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  VAS scale - for subjective assessment of pain intensity, most often in the form of a line with special markings, from 0 - which means complete lack of pain, to 10 - which means unbearable pain (the greatest pain the patient can imagine). On the scale VAS: 0 means no pain, 1-3 mild pain, 4-7 moderate pain, above 7 - severe pain, 10 - unbearable pain.
WHOQOL-BREF | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  WHOQOL-BREF questionnaire for assessing quality of life - which allows for obtaining an assessment of quality of life for the last 14 days in four assessed domains: somatic, psychological, social and environmental. Answers to questions included in the WHOQOL-Bref scale are classified on a five-point scale, with a higher score indicating a better perception of quality of life in a given area. The obtained number of points is converted to a 100-point scale, with a higher score being considered a sign of higher quality of life.
Stroke Quality of Life Scale - (SSQOL) | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Stroke Quality of Life Scale - (SSQOL) is one of the specific tools used to assess quality of life determined by health status after stroke. SSQOL allows for obtaining a profile in the scope of global quality of life from 2 domains - physical and psychosocial and 12 subscales. Each of the SSQOL subscales contains 3 to 6 items - 49 in total. The SSQOL has two sets of answers, which concern the patient's functioning in the past week. They were developed on the basis of a 5-point Likert scale (1.0 - 5.0), where a higher score indicates better functioning in a given area.
Box and Blocks test | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Box and Blocks test to assess the manual dexterity of the hand. The test consists of a wooden box (53.7 cm x 25.4 cm x 8.5 cm) divided into two parts by a partition and 150 blocks (2.5 cm). The test consists of the patient transferring as many blocks as possible from one compartment of the box to another of equal size within 60 seconds. The box should be placed in the patient's midline so that during transfer the blocks are transferred through the partition. Before performing the actual test, the patient can perform the test for 15 seconds and start the test with the unoccupied hand. A higher number of transferred blocks indicates better manual dexterity of the patient.
Franchay scale | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Franchay scale for assessing the grip function of the hand. The scale consists of 7 tasks - pass/fail, and the patient scores 1 point for each successfully completed task or 0 for failure to perform. Using the paretic hand, the patient attempts to unscrew a jar, lift and put back a 2-inch diameter cylinder (later ½ inch diameter). The next task is to use the paretic hand to drink water from a glass, comb one's hair, open and close a clothing case. The maximum possible sum of points for performing the above activities is 7. The more points the patient scores, the better the manual dexterity of the hand. This scale is a measure of proximal control of upper limb movements and manual dexterity of the hand. Studies show that the Franchay scale is characterized by excellent reliability and is a reliable tool in assessing the grip function of the hand of people after stroke
Fugl-Meyer Assessment (FMA) | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Fugl-Meyer Motor Assessment Scale for Upper Extremity for assessing the motor skills of the hand. The hand function test assesses: precision movements and grip. The score is 0-2 for each activity. Items are scored on a 3-point ordinal scale:
  0 = cannot perform
  1. = performs partially
  2. = performs fully. The more points the patient scores, the better the motor skills of the hand.
Hand grip strength | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Pinching strength of the fingers | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
Functional electrostimulation and EMG | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Functional electrostimulation and EMG using the Stella Bio device. This is a muscle activity imaging test. The reading of the bioelectric activity of the muscles is transmitted in the form of numbers and graphs to the screen of the device, thanks to which feedback is obtained on the muscle activity.
Body height | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Body height will be measured to the nearest 0.1 cm using a portable PORTSTAND 210 stadiometer.
Body weight | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Body weight will be measured to the nearest 0.1 kg using a Tanita 780 body composition analyzer
Body mass index (BMI) | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  The body mass index (BMI) will be calculated, and then the BMI value will be related to the obesity classification according to the WHO: ≤ 18.49 underweight, 18.5 - 24.99 normal body weight, 25 - 29.99 overweight, ≥ 30 obesity.
The Modified Ashworth Scale (MAS) | Measurement during the patient's enrolment
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
  0 - No increase in muscle tone
  1 - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 - Considerable increase in muscle tone passive, movement difficult 4 - Affected part(s) rigid in flexion or extension
Assessment of paretic limb function with the Brunnström scale. | Measurement during the patient's enrolment
  Motor performance (function) of extremities is to be assessed using Brunnström scale. This is a six-point scale designed to evaluate performance (function) of paretic extremities.The higher the score, the better. 1-No moves 6-Precise movements, ball throw, button fastening and unfastening
Assessment of disability level, using the modified Rankin scale (MRS) | Measurement during the patient's enrolment
  Assessment of disability using the modified Rankin scale (MRS) Score Description 0 - No symptoms at all 1- No significant disability despite symptoms; able to carry out all usual duties and activities; 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3 - Moderate disability; requiring some help, but able to walk without assistance; 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6 - Dead TOTAL (0-6)
Range of motion of the joints of the upper limbs | First measurement before rehabilitation treatment, second after 3 weeks of rehabilitation program
  Measurement using the R500 goniometer to assess the range of motion of the joints of the upper limbs. The device works with an accuracy of one degree and is automatically transferred to special software via Bluetooth wireless connection.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bylicki, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland